CLINICAL TRIAL: NCT06733207
Title: Comparison of Clinical Pupillary Assessment by Healthcare Professionals With Pupillometry
Brief Title: Pupillometry Use & Professional's Inspection : Leveling Subjectivity
Acronym: PUPILS
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO24112
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Intensive Care; Pupil Assessment; Pupillometry; Neurological Examination; Clinical Competence; Nursing Assessment; Diagnostic Techniques and Procedures; Comparative Effectiveness Research; Interprofessional Relations; Observer Variation
Keywords: Intensive Care; Pupil assessment; Pupillometry; Neurological Examination; Clinical Competence; Nursing Assessment; Diagnostic Techniques and Procedures; Comparative Effectiveness Research; Interprofessional Relations; Observer Variation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in Intensive Care: This prospective diagnostic study involves a single cohort of patients undergoing pupil assessment. Within this cohort, the evaluations will be performed by three distinct sub-cohorts of healthcare providers:
  * Senior physicians : Experienced anesthesiologists or critical care specialists with extensive training in pupil evaluation and neurological assessment.
  * Anesthesiology Residents: Trainees responsible for assessing the pupils of the patients, focusing on their developing assessment skills.
  * Nurses: Registered nurses involved in the assessment of patients' pupils as part of their routine care.
  Interventions: Other: Pupil examination

INTERVENTIONS:
Other: Pupil examination — Pupil assessment : bilateral clinical examination of the patient's pupils, assessed in qualitative data : mydriasis, myosis, pupillary light reflex, anisocoria or isochoria.

SUMMARY:
This prospective, non interventionneal, mono-centric study aims to evaluate the accuracy and quality of pupil assessment among three different groups: senior physicians, anesthesiology residents, and nurses. Pupil assessment is a critical component in anesthesia and emergency medicine, providing essential information about a patient's neurological status and response to medications.

DETAILED DESCRIPTION:
This study aims to assess if there is a significant differences in the accuracy and reliability of pupil evaluations between senior physicians, residents, and nurses when compared to the gold standard of pupillometry, an objective and precise measurement technique.

The study will involve a series of assessments where each participant will evaluate patients' pupils under controlled conditions. The results will be compared against the measurements obtained from pupillometry to determine how closely each group aligns with this standard.

By identifying any discrepancies in pupil assessment skills among the different professional groups, we hope to highlight areas for improvement in training and practice. Ultimately, this research aims to enhance patient care by ensuring that pupil evaluations are performed accurately and consistently across all levels of healthcare providers.

The findings from this study could lead to improved training protocols and potentially influence guidelines for pupil assessment in clinical practice, contributing to better patient outcomes in anesthesia and emergency settings.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in Intensive Care
* Patients who gave their consent to participate to the study, or, if incapable of giving their consent, for whom their designated trusted person has provided their consent.

Exclusion Criteria:

* Aged under 18 years
* Undergoing ocular surgery
* Unable to evaluate both pupils
* Not affiliated with a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized in the Surgical Intensive Care Unit at CHU de Reims who have consented to participate in the study, or for whom a designated trusted person has provided consent for their participation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
pupil examination | Day 1
  comparison of pupil examination through an intraclass correlation coefficient for each category of healthcare professional to measure the concordance between the subjective pupillary examination and pupillometry

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France